CLINICAL TRIAL: NCT01156909
Title: B-lymphocyte Depletion Using the Monoclonal Anti-CD20 Antibody Rituximab in Chronic Fatigue Syndrome. An Open Label Phase II Study With Rituximab Induction and Maintenance Treatment
Brief Title: B-cell Depletion Using the Monoclonal Anti-CD20 Antibody Rituximab in Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/1318
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Chronic fatigue syndrome; CFS; Myalgic encephalomyelitis; Rituximab; B-cell depletion
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): Rituximab induction using two infusions (500mg/m2, max 1000 mg) two weeks apart, followed by maintenance Rituximab infusions (500 mg/m2, max 1000 mg) after 3, 6, 10 and 15 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Two infusions of Rituximab 500 mg/m2 (max 1000 mg) given two weeks apart, followed by maintenance Rituximab infusions 500 mg/m2 (max 1000 mg) at 3, 6, 10, and 15 months.
  Approved amendment: for patients with gradual improvement in CFS/ME symptoms after 12 months follow-up, but not having reached a clear response, up to 6 additional Rituximab infusions (500 mg/m2, max 1000 mg) may be given during the following 12 months period.

SUMMARY:
Based on pilot patient observations, and experience from the prior study KTS-1-2008, the investigators anticipate that chronic fatigue syndrome patients may benefit from B-cell depletion therapy using Rituximab induction with maintenance treatment.

The hypothesis is that at least a subset of CFS patients have an activated immune system involving B-lymphocytes, and that prolonged B-cell depletion may alleviate symptoms.

ELIGIBILITY:
Inclusion Criteria:

* patients with CFS
* age 18-66 years
* informed consent

Exclusion Criteria:

* patients with fatigue, not fulfilling criteria for CFS
* pregnancy or lactation
* previous malignant disease except basal cell carcinoma of skin and cervical carcinoma in situ
* previous major immunological disease, except autoimmune diseases such as diabetes mellitus or thyroiditis
* previous long-term use of immunosuppressive drugs, except steroids e.g. in obstructive lunge disease
* endogenous depression
* lack of ability to comply by the protocol
* multi-allergy with risk of serious drug reaction
* reduced renal function (creatinin > 1.5 x UNL)
* reduced liver function (bilirubin or transaminases > 1.5 x UNL)
* HIV positivity
* evidence of clinically significant infection

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes. | Major response of at least six weeks duration, independent on when occuring, during the follow-up period.
  The primary endpoint is defined as major response of the CFS symptoms, of at least six weeks duration, independent on when during 36 months follow-up the response period(s) occurs. Single such response periods, and the sum of these, are recorded.

SECONDARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes. | At 3, 6, 10, 15, 20, 24, 30, 36 months after intervention
  The secondary outcome measures are effect on the CFS symptoms, by evaluation at 3, 6, 10, 15, 20, 24, 30, and 36 months after first intervention (i.e. first Rituximab infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Mella, PhD, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Department of Oncology, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Fluge O, Mella O. Clinical impact of B-cell depletion with the anti-CD20 antibody rituximab in chronic fatigue syndrome: a preliminary case series. BMC Neurol. 2009 Jul 1;9:28. doi: 10.1186/1471-2377-9-28. PMID 19566965
- [Derived] Fluge O, Risa K, Lunde S, Alme K, Rekeland IG, Sapkota D, Kristoffersen EK, Sorland K, Bruland O, Dahl O, Mella O. B-Lymphocyte Depletion in Myalgic Encephalopathy/ Chronic Fatigue Syndrome. An Open-Label Phase II Study with Rituximab Maintenance Treatment. PLoS One. 2015 Jul 1;10(7):e0129898. doi: 10.1371/journal.pone.0129898. eCollection 2015. PMID 26132314